CLINICAL TRIAL: NCT02075580
Title: Totally Implantable Venous Access Devices (TIVAD): Impact on Quality of Life and Body Image
Brief Title: Totally Implantable Venous Access Devices: Quality of Life and Body Image
Acronym: BI-PORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Fondazione Guido Berlucchi (Other)
Responsible Party: Principal Investigator, Marco Scarpa, MD, PhD, Istituto Oncologico Veneto IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BI-PORT
Record Dates: First submitted 2014-02-05; First posted 2014-03-03 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Neoplasms Undergoing Chemotherapy
Keywords: cancer, quality of life, body-image, subcutaneous-implant
MeSH Terms: conditions — Neoplasms | interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- psychological support (Experimental): Arm A will undergo psychological support and standard care prior and post TIVAD (Totally Implantable Venous Access Devices) insertion Arm B will undergo standard care prior and post TIVAD insertion
  Interventions: Behavioral: psychological support (interactive/cognitive strategies)
- standard care (No Intervention): this arm does not receive psychological support before and after Totally Implantable Venous Access Devices positioning

INTERVENTIONS:
Behavioral: psychological support (interactive/cognitive strategies) — * cognitive/behavioural intervention (6 times starting from hospital admission, in 90 days; for arm of intervention)
  * metacognitive techniques (6 times starting from hospital admission, in 90 days; for arm of intervention)
  * psychoeducational intervention (6 times starting from hospital admission; for arm of intervention)
  * questionnaires: EORTC questionnaires and a written structured interview (3 times: hospital admission,15 days after surgical intervention, 90 days after intervention; in both arms)
  Arms: psychological support

SUMMARY:
Our hypothesis is that totally Implantable Venous Access Devices in neoplastic patients modify body image and self-representation. Therefore, the purpose of this study is to evaluate the efficacy of psychological intervention on patients undergone this surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* neoplastic patients
* adults
* not visible demolitive interventions
* not psychopathological diagnosis
* language understanding

Exclusion Criteria:

* not neoplastic patients
* psychopathological diagnosis
* language misunderstanding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Generic and quality of life and body image | 15 days
  EORTC (European Organization for Research and Treatment of Cancer) questionnaire:
  BR23 (Breast questionnaire, used just for BI scale, that is Body Image items)

SECONDARY OUTCOMES:
Satisfaction with care | 15 days
  EORTC (European Organization for Research and Treatment of Cancer) questionnaire: QLQ C30 (Quality of Life Questionnaire)

OTHER OUTCOMES:
Generic and quality of life and body image | 15 days
  textual analysis of discoursive modalities used by patient in self-description
Generic and quality of life and body image | 15 days
  EORTC questionnaire: IN-PATSAT32 (patient satisfaction questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Veneto Institute of Oncology IOV-IRCCS, Padua, Italy

REFERENCES:
- [Derived] Pinto E, Granziera E, Cagol M, Cappellato S, Alfieri R, Mari V, Meroni M, Zagonel V, Conte P, Pilati P, Castoro C, Cavallin F, Scarpa M. Totally Implantable Venous Access Devices: A Randomized Controlled Trial on the Effect of Psychological Support on Quality of Life and Body Image (BI-PORT). Front Psychol. 2021 Nov 12;12:703497. doi: 10.3389/fpsyg.2021.703497. eCollection 2021. PMID 34867586